CLINICAL TRIAL: NCT00412893
Title: A Phase III, Double Blind, Randomized Study to Evaluate Safety and Efficacy of BAL8557 Versus Voriconazole for Primary Treatment of Invasive Fungal Disease Caused by Aspergillus Species or Other Filamentous Fungi.
Brief Title: Isavuconazole (BAL8557) for Primary Treatment of Invasive Aspergillosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9766-CL-0104; WSA-CS-004 (Other: Basilea Protocol ID); 2006-003868-59 (EudraCT Number)
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Aspergillosis; Invasive Fungal Infection
Keywords: Invasive fungal disease; BAL8557; Isavuconazole; ASP9766; Filamentous fungi; Phase III; Aspergillus species
MeSH Terms: conditions — Aspergillosis; Invasive Fungal Infections | interventions — isavuconazole; Voriconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isavuconazole (Experimental): Participants received a loading dose of isavuconazole, 200 mg three times a day by intravenous infusion (IV) for the first 2 days followed by a maintenance dose from Day 3 of 200 mg once daily either IV or orally until they reached a treatment endpoint or for a maximum of 84 days.
  Interventions: Drug: Isavuconazole
- Voriconazole (Active Comparator): Participants received a loading dose of voriconazole, 6 mg/kg every 12 hours IV for the first 24 hours, followed by a maintenance dose of 4 mg/kg every 12 hours by IV on Day 2. Beginning on Day 3, participants received 4 mg/kg every 12 hours by IV or 200 mg every 12 hours orally, until they reached a treatment endpoint or for a maximum of 84 days.
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Isavuconazole — Loading doses were administered as IV infusion and maintenance doses were administered as IV infusion or oral (capsules).
  Other Names: ASP9766; BAL8557
  Arms: Isavuconazole
Drug: Voriconazole — Loading doses were administered as IV infusion and maintenance doses were administered as IV infusion or oral (capsules).
  Other Names: VFend
  Arms: Voriconazole

SUMMARY:
The purpose of this study is to compare the efficacy and safety of isavuconazole versus voriconazole in the treatment of patients with invasive aspergillosis.

DETAILED DESCRIPTION:
Acute invasive fungal infections caused by aspergillus, zygomycetes and other filamentous fungi remain life threatening diseases. Early treatment with highly effective anti-fungals reduces mortality. This study investigates the efficacy and safety of isavuconazole in the treatment of invasive fungal diseases, caused by Aspergillus or other filamentous fungi.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have proven, probable or possible invasive fungal disease caused by Aspergillus species or other filamentous fungi
* Female patients must be non-lactating and at no risk for pregnancy

Exclusion Criteria:

* Patients with invasive fungal infections other than Aspergillus species or other filamentous fungi
* Evidence of hepatic dysfunction at Baseline or moderate to severe renal dysfunction
* Patients with chronic aspergillosis, or aspergilloma or allergic bronchopulmonary aspergillosis
* Patients who have received more than 4 days of systemic antifungal therapy other than fluconazole within the 7 days prior to the first administration of study medication
* Patients previously enrolled in a Phase III study with isavuconazole
* Patients with a body weight </= 40 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2007-03-07 (Actual); Primary Completion 2013-03-28 (Actual); Study Completion 2013-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (103):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - University of California at San Francisco, San Francisco, California
  - University of Chicago, Division of Infectious Diseases, Chicago, Illinois
  - Indiana BMT, Springfield, Illinois
  - Springfield Clinic LLP, Springfield, Illinois
  - Infectious Disease of Indiana, Indianapolis, Indiana
  - Brigham & Womens Hospital, Boston, Massachusetts
  - Worcester, Massachusetts
  - Upstate Infectious Diseases Association LLP, Albany, New York
  - Regional Infection Diseases Infusion Center Inc., Lima, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Argentina (4):
  - Buenos Aires
  - Capital Federal
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma
- Australia (3):
  - Perth
  - Mater Medical Centre, South Brisbane
  - Woolloongabba
- Belgium (5):
  - AZ ST Jan, Bruges
  - Institut Jules Bordet, Brussels
  - ULB Hospital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (5):
  - Felicio Rocho, Belo Horizonte
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Hospital das Clinicas da UFPR, Curitiba
  - Hospital de Clinicas da FMUSP - Ribeirao Preto, Ribeirão Preto
  - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro
- Canada (2):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Hamilton Health Sciences - Henderson Site, Hamilton
- Chile (3):
  - Santiago
  - Hospital Dr. Hernan Henriquez Aravena, Temuco
  - Valdivia
- China (12):
  - 3rd Hospital, Peking University, Beijing
  - The 1st Hospital, Jilin University, Changchun
  - The Third Xiangya Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - The Affiliated Union Hospital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital, Med. School, Zhejiang Uni., Hangzhou
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - The 1st Affiliated Hospital of Guangxi Medical University, Nanning
  - Huashan Hospital, Insitute of Antibiotics, Shanghai
  - No.6 Renmin Hosp. of Shanghai City, Shanghai
  - Chang Hai Hospital, Shanghai
  - Wuhan Union Hospital, Wuhan
- Egypt (3):
  - Alexandria University Hospital, Alexandria
  - National Cancer Institute, Cairo
  - Nasser Institute, Cairo
- France (5):
  - Dijon
  - CHU de Nantes - Hôpital Hôtel Dieu, Nantes
  - Hotel Dieu, Nantes
  - Hôpital Hautepierre, Strasbourg
  - Hôpital de brabois adultes, Vandœuvre-lès-Nancy
- Germany (7):
  - Universitaetsklinikum Aachen, Aachen
  - Charité Universitaetsmedizin Berlin- Campus Charité Mitte, Berlin
  - Universitaet Koeln, Cologne
  - Universitaetsklinik Leipzig, Leipzig
  - Lübeck
  - Klinikum Schwabing, München
  - Medizinische klinik und Polyklinik II, Würzburg
- Hungary (3):
  - Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Szegedi Tudomanyegyetem, Szeged
- India (8):
  - Apollo Hospitals, Hyderabad, Andh Prad
  - Sterling Hospital, Ahmedabad, Gujarat
  - Kasturba Medical College and Hospital, Mangalore, Karna
  - Shirdi Sai Baba Cancer Hospital K. M. C. Hospital, Manipal, Karna
  - Tata Memorial Hopital, Department of Anesthesia, Mumbai, Mahara
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Mahara
  - Sahyadri Hospital, Pune, Mahara
  - Noida, Uttar Prad
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah Universtiy Hospital - Ein Kerem, Jerusalem
  - Rabin MC, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky MC Ichilov Hospital Tel Aviv, Tel Aviv
- Italy (2):
  - Unità Funzionale di Ematologia; Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
- Kuala Lumpur, Malaysia
- Mexico (2):
  - México
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Nijmegen, Netherlands
- Palmerston North, New Zealand
- Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw, Poland
- Russia (5):
  - State Institution "Hematology Research Center" RAMS, Moscow
  - Republican Hospital named after V.A. Baranov, Petrozavodsk
  - Leningrad Regional Hospital, Saint Petersburg
  - St-Petersburg MA Postgraduate Education, Saint Petersburg
  - Saint Petersburg
- South Korea (5):
  - Gachon University Gil Hospital, Incheon
  - Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
- Salamanca, Spain
- Zurich, Switzerland
- Thailand (6):
  - Songklanagarind Hospital, Hat Yai
  - Khon Kaen
  - Maharat Nakhon Ratchasima Hospital, Muang
  - Srinagarind Hospital, Muang
  - Maharaj Nakorn Chiang Mai Hospital, Muang
  - Songkhla
- Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Hamed K, Engelhardt M, Kovanda LL, Huang JJ, Yan J, Aram JA. Post-hoc analysis of the safety and efficacy of isavuconazole in older patients with invasive fungal disease from the VITAL and SECURE studies. Sci Rep. 2023 Apr 25;13(1):6730. doi: 10.1038/s41598-023-31788-1. PMID 37185921
- [Derived] Kovanda LL, Kolamunnage-Dona R, Neely M, Maertens J, Lee M, Hope WW. Pharmacodynamics of Isavuconazole for Invasive Mold Disease: Role of Galactomannan for Real-Time Monitoring of Therapeutic Response. Clin Infect Dis. 2017 Jun 1;64(11):1557-1563. doi: 10.1093/cid/cix198. PMID 28472247
- [Derived] Maertens JA, Raad II, Marr KA, Patterson TF, Kontoyiannis DP, Cornely OA, Bow EJ, Rahav G, Neofytos D, Aoun M, Baddley JW, Giladi M, Heinz WJ, Herbrecht R, Hope W, Karthaus M, Lee DG, Lortholary O, Morrison VA, Oren I, Selleslag D, Shoham S, Thompson GR 3rd, Lee M, Maher RM, Schmitt-Hoffmann AH, Zeiher B, Ullmann AJ. Isavuconazole versus voriconazole for primary treatment of invasive mould disease caused by Aspergillus and other filamentous fungi (SECURE): a phase 3, randomised-controlled, non-inferiority trial. Lancet. 2016 Feb 20;387(10020):760-9. doi: 10.1016/S0140-6736(15)01159-9. Epub 2015 Dec 10. PMID 26684607
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=52

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consenting adult patients with proven, probable or possible invasive fungal disease (IFD) caused by Aspergillus species or other filamentous fungi, meeting the inclusion/exclusion criteria, were enrolled in the study.
Pre-assignment Details: Participants were stratified by geographic location (North America; Western Europe plus Australia and New Zealand; and Other Regions), whether or not they underwent an allogeneic bone marrow transplant (BMT) and whether or not they had uncontrolled malignancy.
Period: Overall Study
Arm/Group | Isavuconazole | Voriconazole
Started | 263 | 264
Received Treatment | 258 (One participant randomized to this group received voriconazole treatment for the first 7 days) | 258
Completed | 118 (Defined as completed treatment) | 120 (Defined as completed treatment)
Not Completed | 145 | 144
Not completed — Adverse Event | 31 | 53
Not completed — Death | 17 | 21
Not completed — Insufficient Therapeutic Response | 39 | 23
Not completed — Lost to Follow-up | 2 | 1
Not completed — Violation of Selection at Entry | 17 | 10
Not completed — Other Protocol Violation | 10 | 6
Not completed — Did Not Cooperate | 12 | 9
Not completed — Administrative Reason | 12 | 15
Not completed — Randomized but Never Received Study Drug | 5 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted of all randomized participants who received at least one administration of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Isavuconazole | Voriconazole | Total
Number analyzed (Participants) | 258 | 258 | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (16.15) | 51.2 (15.85) | 51.1 (15.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 95 | 208
  Male | 145 | 163 | 308
Race/Ethnicity, Customized [Number; unit: participants]
  White | 211 | 191 | 402
  Black or African American | 1 | 1 | 2
  Asian | 45 | 64 | 109
  Other | 1 | 1 | 2
  Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 22 | 9 | 31
  Not Hispanic or Latino | 236 | 248 | 484
  Missing | 0 | 1 | 1
Hematologic Malignancy Status [Number; unit: participants]
  Yes | 211 | 222 | 433
  No | 47 | 36 | 83
Prior Allogeneic Bone Marrow Transplant (BMT) [Number; unit: participants] — Allogeneic BMT Status was defined as Yes for patients indicated as having a BMT, hematopoietic stem cell transplant (HSCT) or other progenitor cell transplant with type of transplant identified as allogeneic.
  participants
    Yes | 54 | 51 | 105
    No | 204 | 207 | 411
Uncontrolled Malignancy Status [Number; unit: participants] — Uncontrolled malignancy was defined as participants who per Investigator judgment had active malignancy (new diagnosis or relapse).
  participants
    Yes | 173 | 187 | 360
    No | 85 | 71 | 156
Neutropenic Status [Number; unit: participants] — The presence or absence of neutropenia was defined as an absolute neutrophil count (ANC) < 0.5 x 10^9/L (< 500/mm^3).
  participants
    Yes | 163 | 175 | 338
    No | 95 | 83 | 178

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Through Day 42
Description: All-cause mortality is represented as the percentage of participants who died after first dose of study drug through Day 42 from any cause. Participants with unknown survival status through Day 42 were included as deaths in the calculation.
Time Frame: Through Day 42
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 258 | 258
percentage of participants | 18.6 | 20.2
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; Approximately 255 patients per group were to be enrolled to ensure at least 80% power to demonstrate that the upper bound of the 95% confidence interval (CI) for a treatment difference in favor of the comparator was no larger than 10%; Test type: Non-Inferiority or Equivalence — The upper bound of the 95% CI for the treatment difference was compared to the protocol prespecified non-inferiority margin of 10%. If the upper bound was smaller than 10%, isavuconazole was declared as non-inferior to voriconazole with respect to the primary outcome measure; Adjusted Treatment Difference = -1.0, 95% CI 2-sided [-7.759 to 5.683] — The treatment difference (isavuconazole minus voriconazole) was calculated using a stratified Cochran-Mantel-Haenszel (CMH) method. The strata included Geographical Regions, Allogeneic BMT Status and Uncontrolled Malignancy Status

2. Secondary Outcome: Percentage of Participants With an Overall Outcome of Success Evaluated by the Data Review Committee (DRC)
Description: The DRC was an independent, blinded committee consisting of experts in the field of infectious disease who assessed patients' outcomes. The overall response was based on the DRC-assessed clinical, mycological and radiological responses. Success was defined as the resolution or partial resolution of all attributable clinical symptoms and physical findings, the eradication or presumed eradication of the original causative organism cultured or identified by histology/cytology at Baseline and a > 50% improvement in radiological response from Baseline (or improvement of at least 25% from Baseline for the Day 42 analysis or End of Treatment if it occurred prior to Day 42). End of treatment (EOT) is the last day of study drug administration. For the Day 42 and Day 84 analyses, any visits that the DRC assessed as Not Done were considered a failure for that visit. A death before Day 42 was also considered a failure, even if the DRC assessed the participant to be a success prior to death.
Time Frame: Day 42, Day 84 and End of Treatment. The median duration of study drug administration was 45 days.
Population: Modified Intent-to-treat (mITT) population consisted of ITT participants who had proven or probable IFD as determined by the DRC.
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 143 | 129
percentage of participants
  Day 42 | 35.7 | 35.7
  Day 84 | 25.2 | 32.6
  End of Treatment | 35.0 | 36.4
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; End of Treatment comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 1.6, 95% CI 2-sided [-9.336 to 12.572] — The adjusted treatment difference (Voriconazole-Isavuconazole) was calculated by a stratified CMH method with the strata of Geographical Region, Allogeneic BMT Status and Uncontrolled Malignancy Status
Statistical Analysis 2: Comparison: Isavuconazole vs Voriconazole; Day 42 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = -0.5, 95% CI 2-sided [-11.277 to 10.329] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Isavuconazole vs Voriconazole; Day 84 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 8.2, 95% CI 2-sided [-1.993 to 18.379] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: All-cause Mortality Through Day 84
Description: All-cause mortality is represented as the percentage of participants who died after first dose of study drug through Day 84 from any cause. Participants with unknown survival status through Day 84 were included as deaths in the calculation.
Time Frame: Through Day 84
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 258 | 258
percentage of participants | 29.1 | 31.0
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; Test type: Superiority or Other; Adjusted Treatment Difference = -1.4, 95% CI 2-sided [-9.150 to 6.340] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With an Overall Outcome of Success Evaluated by Investigator
Description: Overall response based on investigators' assessments was not derived as it was not deemed necessary because participants overall response status was determined by the DRC. All investigators' assessments of clinical, mycological and radiological responses are analyzed separately (see Outcome Measures 8-10).
Time Frame: Day 42, Day 84 and End of Treatment. The median duration of study drug administration was 45 days.
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With a Clinical Response Assessed by the DRC
Description: Blinded assessments of clinical symptoms and physical findings of invasive fungal disease were performed by the independent DRC. Clinical response is defined as the resolution or partial resolution of all attributable clinical symptoms and physical findings. Failure is defined as no resolution of any attributable clinical symptoms and physical findings and/or worsening. Participants with no attributable signs and symptoms present at Baseline and no symptoms attributable to invasive fungal disease (IFD) developed post-baseline were classified as "Not Applicable." End of treatment is the last day of study drug administration.
Time Frame: Day 42, Day 84 and End of Treatment. The median duration of study drug administration was 45 days.
Population: Modified intent-to-treat population. Any visits the DRC assessed as not done were considered as missing and included as a failure; participants with a Not Applicable assessment were excluded. The number of participants included in the analysis at each time point in indicated by "n".
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 143 | 129
percentage of participants
  Day 42 (n=139, 120) | 64.0 | 57.5
  Day 84 (n=141, 124) | 46.1 | 44.4
  End of Treatment (n=137, 121) | 62.0 | 60.3
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; End of Treatment Comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 0.4, 95% CI 2-sided [-10.640 to 11.531] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Isavuconazole vs Voriconazole; Day 42 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = -5.8, 95% CI 2-sided [-17.368 to 5.802] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Isavuconazole vs Voriconazole; Day 84 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 0.3, 95% CI 2-sided [-11.116 to 11.758] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Participants With a Mycological Response Assessed by the DRC
Description: Blinded mycological assessments of the participant's invasive fungal disease status were performed by the independent DRC using the results from fungal culture and isolation and/or histology/cytology of biopsy or biological fluid samples from the infected site. Mycological response is defined as eradication or presumed eradication of the original causative organism cultured or identified by histology/cytology at Baseline. Failure was defined as persistence or presumed persistence. Participants with no mycological evidence available at Baseline were classified as "Not Applicable". End of treatment is the last day of study drug administration.
Time Frame: Day 42, Day 84 and End of Treatment. The median duration of study drug administration was 45 days.
Population: Modified intent-to-treat population. Any visits the DRC assessed as not done were considered as missing and included as a failure; participants with a Not Applicable assessment were excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 143 | 129
percentage of participants
  Day 42 | 39.9 | 39.5
  Day 84 | 28.0 | 36.4
  End of Treatment | 37.8 | 41.1
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; End of Treatment comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 3.8, 95% CI 2-sided [-7.429 to 15.087] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Isavuconazole vs Voriconazole; Day 42 Comparison; Test type: Superiority or Other; Adjusted Treatment Difference = -0.7, 95% CI 2-sided [-11.917 to 10.586] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Isavuconazole vs Voriconazole; Day 84 Comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 9.1, 95% CI 2-sided [-1.624 to 19.830] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Percentage of Participants With a Radiological Response Assessed by the DRC
Description: Independent reviews of radiology assessments were completed by radiology experts which were provided to the independent, blinded DRC. Blinded radiological assessments were performed by the DRC. Radiological response is defined as a ≥ 50% improvement from Baseline, or improvement of at least 25% from Baseline for the Day 42 analysis or if end of treatment occurred before Day 42. Participants without any radiology at Baseline were considered "Not Applicable." End of Treatment is the last day of study drug administration.
Time Frame: Day 42, Day 84 and End of Treatment. The median duration of study drug administration was 45 days.
Population: Modified intent-to-treat population. A participant with no post-baseline radiology data with evidence of radiologic disease at Baseline was considered a failure. Participants with a Not Applicable assessment were excluded. The number of participants included in the analysis at each time point is indicated by "n".
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 143 | 129
percentage of participants
  Day 42 (n=141, 128) | 28.4 | 34.4
  Day 84 (n=141, 128) | 22.0 | 29.7
  End of Treatment (n=141, 127) | 29.1 | 33.1
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; End of Treatment comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 5.7, 95% CI 2-sided [-4.936 to 16.268] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Isavuconazole vs Voriconazole; Day 42 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 5.3, 95% CI 2-sided [-5.338 to 16.032] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Isavuconazole vs Voriconazole; Day 84 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 9.0, 95% CI 2-sided [-1.231 to 19.186] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Percentage of Participants With a Clinical Response Assessed by the Investigator
Description: Assessment of clinical symptoms and physical findings of invasive fungal disease were performed by the investigator. Clinical response is defined as the resolution or partial resolution of all attributable clinical symptoms and physical findings. Failure is defined as no resolution of any attributable clinical symptoms and physical findings and/or worsening, or if results were unavailable or the participant was unevaluable. Participants with no attributable signs and symptoms present at Baseline were classified as "Not Applicable." End of treatment is the last day of study drug administration.
Time Frame: Day 42, Day 84 and End of Treatment. The median duration of study drug administration was 45 days.
Population: Modified intent-to-treat population. Missing data for any participant at any visit was included as a failure; participants with a Not Applicable assessment were excluded. The number of participants included in the analysis at each time point in indicated by "n".
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 143 | 129
percentage of participants
  Day 42 (n=137, 120) | 64.2 | 61.7
  Day 84 (n=140, 122) | 41.4 | 44.3
  End of Treatment (n=137, 121) | 62.0 | 64.5
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; End of Treatment comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 5.0, 95% CI 2-sided [-6.043 to 16.026] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Isavuconazole; Day 42 comparison; Test type: Superiority or Other; Adjusted treatment Difference = 0.2, 95% CI 2-sided [-10.873 to 11.220] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Isavuconazole vs Voriconazole; Day 84 comparison; Test type: Superiority or Other; Adjusted treatment Difference = 4.7, 95% CI 2-sided [-6.533 to 15.939] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Percentage of Participants With a Mycological Response Assessed by the Investigator
Description: Mycological assessments of the participant's invasive fungal disease status were performed by the investigator using the results from fungal culture and isolation and/or histology/cytology of biopsy or biological fluid samples from the infected site. Mycological response is defined as eradication or presumed eradication of the original causative organism cultured or identified by histology/cytology at Baseline. Failure was defined as persistence or presumed persistence. Participants with no mycological evidence available at Baseline, or no mycological follow-up results available or indeterminate results were classified as "Not Applicable". End of treatment is the last day of study drug administration.
Time Frame: Day 42, Day 84 and End of Treatment. The median duration of study drug administration was 45 days.
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 143 | 129
percentage of participants
  Day 42 (n=109, 100) | 52.3 | 50.0
  Day 84 (n=126, 117) | 35.7 | 37.6
  End of Treatment (n=107, 100) | 50.5 | 55.0
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; End of Treatment comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 4.4, 95% CI 2-sided [-8.429 to 17.218] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Isavuconazole vs Voriconazole; Day 42 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = -2.5, 95% CI 2-sided [-15.071 to 10.073] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Isavuconazole vs Voriconazole; Day 84 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 2.9, 95% CI 2-sided [-8.633 to 14.499] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Percentage of Participants With a Radiological Response Assessed by the Investigator
Description: Radiological assessments were performed by the investigator. Radiological response is defined as a ≥ 50% improvement from Baseline, or improvement of at least 25% from Baseline for the Day 42 analysis or if end of treatment occurred before Day 42. Failure is defined as a < 25% improvement at any time or results not available. Participants with no signs on radiological images at Baseline were considered "Not Applicable." End of Treatment is the last day of study drug administration.
Time Frame: Day 42, Day 84 and End of Treatment. The median duration of study drug administration was 45 days.
Population: Modified intent-to-treat population. Missing data for any participant at any visit was included as a failure. Participants with a Not Applicable assessment were excluded. The number of participants included in the analysis at each time point is indicated by "n".
Measure: Number; unit: percentage of participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 143 | 129
percentage of participants
  Day 42 (n=142, 128) | 45.1 | 51.6
  Day 84 (n=141, 128) | 38.3 | 41.4
  End of Treatment (n=141, 128) | 43.3 | 47.7
Statistical Analysis 1: Comparison: Isavuconazole vs Voriconazole; End of Treatment comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 6.3, 95% CI 2-sided [-5.145 to 17.696] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Isavuconazole vs Voriconazole; Day 42 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 8.0, 95% CI 2-sided [-3.335 to 19.356] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Isavuconazole vs Voriconazole; Day 84 comparison; Test type: Superiority or Other; Adjusted Treatment Difference = 5.1, 95% CI 2-sided [-6.187 to 16.332] — [estimate comment as in outcome 2, analysis 1]

11. Secondary Outcome: Number of Participants With Adverse Events, Reported by System Organ Class
Time Frame: From the first study drug administration until 28 days after the last dose of study drug. The median duration of study drug administration was 45 days.
Population: The safety analysis set consists of all randomized patients who received at least one dose of study drug according to the study drug that the participant actually received as the first dose. One participant was randomized to isavuconazole but received voriconazole treatment for the first 7 days and is included in the voriconazole arm for safety.
Measure: Number; unit: participants
Arm/Group | Isavuconazole | Voriconazole
Number analyzed (Participants) | 257 | 259
participants
  Patients with ≥ 1 TEAE | 247 | 255
  Gastrointestinal Disorders | 174 | 180
  Infections and Infestations | 152 | 158
  General Disorders / Administration Site Conditions | 148 | 144
  Respiratory, Thoracic and Mediastinal Disorders | 143 | 147
  Metabolism and Nutrition Disorders | 108 | 121
  Nervous System Disorders | 95 | 89
  Skin and Subcutaneous Tissue Disorders | 86 | 110
  Investigations | 85 | 96
  Blood and Lymphatic System Disorders | 77 | 82
  Psychiatric Disorders | 70 | 86
  Musculoskeletal and Connective Tissue Disorders | 69 | 77
  Vascular Disorders | 67 | 77
  Renal and Urinary Disorders | 55 | 58
  Cardiac Disorders | 43 | 57
  Eye Disorders | 39 | 69
  Injury, Poisoning and Procedural Complications | 33 | 39
  Hepatobiliary Disorders | 23 | 42
  Immune System Disorders | 20 | 25
  Neoplasms benign, malignant and unspecified | 19 | 31
  Ear and Labyrinth Disorders | 14 | 13
  Reproductive System and Breast Disorders | 8 | 13
  Endocrine Disorders | 5 | 3
  Congenital, Familial and Genetic Disorders | 3 | 2
  Social Circumstances | 0 | 1

ADVERSE EVENTS:
Time Frame: From the first study drug administration until 28 days after the last dose of study drug. The median duration of study drug administration was 45 days.
Description: The safety analysis set consists of all randomized patients who received at least one dose of study drug according to the study drug that the participant actually received as the first dose. One participant was randomized to isavuconazole but received voriconazole treatment for the first 7 days and is included in the voriconazole arm for safety.
Arm/Group | Isavuconazole | Voriconazole
Serious Adverse Events (participants affected / at risk) | 134/257 | 149/259
Other Adverse Events (participants affected / at risk) | 227/257 | 228/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Isavuconazole (N=257) | Voriconazole (N=259)
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 5
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Pancytopenia (Blood and lymphatic system disorders) | 4 | 3
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 5
Cardio-respiratory arrest (Cardiac disorders) | 2 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Blindness unilateral (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1
Optic neuropathy (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 7
Pyrexia (General disorders) | 8 | 10
Sudden cardiac death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Acute graft versus host disease (Immune system disorders) | 1 | 1
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 2
Acute graft versus host disease in liver (Immune system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 2
Anaphylactic shock (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 4 | 3
Bacteraemia (Infections and infestations) | 0 | 2
Bacterial sepsis (Infections and infestations) | 0 | 4
Bronchitis pneumococcal (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Cerebral aspergillosis (Infections and infestations) | 1 | 0
Clostridium bacteraemia (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 2
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Encephalitis herpes (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 3 | 3
Fusarium infection (Infections and infestations) | 1 | 0
Gastric ulcer helicobacter (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Infusion site infection (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 2
Mucormycosis (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 10
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia moraxella (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 8
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 14 | 10
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 3
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Stenotrophomonas sepsis (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Accident at home (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Burkitt's leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Primary effusion lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Brain stem stroke (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 2 | 1
Febrile convulsion (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 2 | 0
Stupor (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 2
Renal failure acute (Renal and urinary disorders) | 6 | 8
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Isavuconazole (N=257) | Voriconazole (N=259)
Anaemia (Blood and lymphatic system disorders) | 11 | 22
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 22
Tachycardia (Cardiac disorders) | 12 | 21
Visual impairment (Eye disorders) | 4 | 19
Abdominal pain (Gastrointestinal disorders) | 24 | 36
Abdominal pain upper (Gastrointestinal disorders) | 15 | 25
Constipation (Gastrointestinal disorders) | 35 | 54
Diarrhoea (Gastrointestinal disorders) | 59 | 59
Dyspepsia (Gastrointestinal disorders) | 15 | 13
Nausea (Gastrointestinal disorders) | 70 | 78
Vomiting (Gastrointestinal disorders) | 64 | 73
Asthenia (General disorders) | 15 | 20
Chills (General disorders) | 27 | 22
Fatigue (General disorders) | 27 | 18
Mucosal inflammation (General disorders) | 23 | 14
Oedema (General disorders) | 13 | 18
Oedema peripheral (General disorders) | 26 | 31
Pyrexia (General disorders) | 53 | 72
Cytomegalovirus infection (Infections and infestations) | 15 | 21
Oral herpes (Infections and infestations) | 13 | 14
Alanine aminotransferase increased (Investigations) | 13 | 17
Aspartate aminotransferase increased (Investigations) | 11 | 14
Blood alkaline phosphatase increased (Investigations) | 12 | 14
Gamma-glutamyltransferase increased (Investigations) | 16 | 22
Decreased appetite (Metabolism and nutrition disorders) | 22 | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 45 | 55
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 15
Dizziness (Nervous system disorders) | 10 | 14
Headache (Nervous system disorders) | 40 | 38
Anxiety (Psychiatric disorders) | 20 | 17
Confusional state (Psychiatric disorders) | 16 | 19
Insomnia (Psychiatric disorders) | 23 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 28
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 25
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 14 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Rales (Respiratory, thoracic and mediastinal disorders) | 5 | 14
Erythema (Skin and subcutaneous tissue disorders) | 9 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 15
Rash (Skin and subcutaneous tissue disorders) | 17 | 26
Hypertension (Vascular disorders) | 25 | 31
Hypotension (Vascular disorders) | 20 | 26

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication for review and comment. Sponsor may delay the publication for up to 60 days to seek patent protection.